CLINICAL TRIAL: NCT04697914
Title: The Effect of a Discharge Sock Model in General and Thermal Comfort and Plantar Pressures: Randomized Controlled Trial.
Brief Title: The Effect of a Discharge Sock Model in Comfort: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Alfonso Martínez Nova, Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INDIGO
Record Dates: First submitted 2020-12-16; First posted 2021-01-06 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Foot Diseases; Metatarsalgia; Pain
Keywords: foot; metatarsalgia; pain; pressure relief; socks; confort
MeSH Terms: conditions — Foot Diseases; Metatarsalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Sock (Placebo Comparator): Control comercial Socks (Lurbel Tierra). These socks are designed to perform trekking.
  Interventions: Diagnostic Test: Plantar pressures will be measured in 7 zones using the Footscan® platform following the two-step method. Three plantar pressures measurements were made for each foot.
- Experimental Relief Pressure sock (Experimental): Experimental Socks (Lurbel Tierra based), with a discharge element (in the own fabric and fibres of the sock).
  Interventions: Diagnostic Test: Plantar pressures will be measured in 7 zones using the Footscan® platform following the two-step method. Three plantar pressures measurements were made for each foot.

INTERVENTIONS:
Diagnostic Test: Plantar pressures will be measured in 7 zones using the Footscan® platform following the two-step method. Three plantar pressures measurements were made for each foot. — to protect the metatarsus and prevent the appearance of foot pain.
  Other Names: Thermal picture. An infrared camera (Flir e60bx) will measure skin temperature. This study mapped out five subregions of anatomic interest over the foot.; Confort survey. An standardized confort survey about different issues of the socks will be fulfilled before and after walking.

SUMMARY:
Metatarsalgia is a common set of symptoms in the forefoot, characterized by pain under one or more metatarsal heads. The invention of a utility model, the U202030700, designed by the study's principal investigator aims to protect the metatarsus and prevent the appearance of foot pain.

The hypothesis of this research project is based on the fact that using our proposed sock with metatarsal discharge plate will bring advantages in terms of pain reduction, increased comfort, temperature reduction and change in plantar pressures received in the second and third metatarsals joint area versus the use of control socks (without discharge plate).

Participants will be subjects with pain in the plantar metatarsal area that will answer few questions and a podiatric exam to determine if meet the study requirements and then a plantar pressures, foot temperature and confort wit the two kind of socks will be taken.

Confort survey, thermal pictures and plantar pressures will be taken (in first term) before and after a brief walk (5 to 10 minutes) and in a second experiment (second term) after a long walk (more than 1 hour).

DETAILED DESCRIPTION:
Metatarsalgia is a common set of symptoms in the forefoot, characterized by pain under one or more metatarsal heads. First option should opt for conservative treatments, among these it is noteworthy the application of pressure relief elements from these anatomical zones. These elements, usually made of soft materials such as felt or foams of different compositions, are arranged covering the entire metatarsal area, with the exception of the compromised sector, that is, overloaded and painful, giving rise to discharge elements with a geometry similar to a U. In this way, the other areas of the metatarsus support the discharge element leaving exposed the overloaded area, so that it reduces or avoids its direct support on the support surface, thus mitigating the excess pressure in the compromised area and therefore, pain.. It is therefore desirable to have unloading elements of the metatarsal area, easy to use by a user and that do not involve major alterations in their usual clothing.

Different types of socks are known with configurations which give them beneficial effects on health. However, these existing models have not specifically focused on the plantar part of the sock, there is therefore no simple and economical solution for the protection of the metatarsus and the mitigation of pain and discomfort usually caused by its pathologies. This has been solved by the invention of a utility model, the U202030700, designed by the study's principal investigator and his research group.

The hypothesis of this research project is based on the fact that using our proposed sock with metatarsal discharge plate will bring advantages in terms of pain reduction, increased comfort, temperature reduction and change in plantar pressures received in the second and third metatarsals joint area versus the use of control socks (without discharge plate).

Specific objectives:

- To record the differences of plantar pressures, thermal and general confort with control socks and experimental socks after a briefs walks.

The type of intervention will be randomly assigned, meaning neither participant nor the secondary researchers knows the sock worn. The principal investigator (Alfonso Martínez Nova) will perform the randomization.

Participants. Subjects with pain in the plantar metatarsal area are suitable to participate in the study.

Participants will answer few questions and a podiatric exam to determine if meet the study requirements and then:

Answering a survey on health status and pain in the metatarsal area mainly. Collection of the necessary data (plantar pressures, foot temperature and confort wit the two kind of socks.

Materials: Experiment socks and control (same fiber, fabric, weight). Pressure platform Footscan. Flir e60bx thermographic camera.

Confort survey, thermal pictures and plantar pressures will be taken (in first term) before and after a brief walk (5 to 10 minutes) and in second term, before and after a long walk (more than 1 hour).

The new sock aimed to protect the metatarsus and prevent the appearance of foot pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with mild discomfort in the plantar metatarsal area of the foot

Exclusion Criteria:

* Subjects with severe disorders of the foot, gait impairment, foot deformations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in plantar pressures measurements. | 10 minutes (first experiment) and more than 1 hour (second experiment)
  Plantar pressures will be measured in 7 zones using the Footscan® platform following the two-step method. Three plantar pressures measurements were made for each foot.
Change from Baseline in plantar temperature measurements. | 10 minutes (first experiment) and more than 1 hour (second experiment)
  An infrared camera (Flir e60bx) will measure skin temperature. This study mapped out five subregions of anatomic interest over the foot.
Change from Baseline foot confort wearing socks. | 10 minutes (first experiment) and more than 1 hour (second experiment)
  An standardized confort survey about different issues of the socks will be fulfilled before and after walking.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Martínez Nova, PhD, Principal Investigator — University of Extremadura
Locations (1):
- Alfonso Martínez Nova, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Nova A, Jimenez-Cano VM, Caracuel-Lopez JM, Gomez-Martin B, Escamilla-Martinez E, Sanchez-Rodriguez R. Effectiveness of a Central Discharge Element Sock for Plantar Temperature Reduction and Improving Comfort. Int J Environ Res Public Health. 2021 Jun 3;18(11):6011. doi: 10.3390/ijerph18116011. PMID 34205056